CLINICAL TRIAL: NCT01664702
Title: Substrate Oxidation in Children in Response to Exercise With High and Low Dairy Intake
Brief Title: Substrate Oxidation in Children in Response to High and Low Dairy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSCL15253; DMI1096 (Other Grant/Funding Number: Dairy Management Inc.)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Childhood Obesity
Keywords: Dairy; obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Dairy Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recommended dairy diet (Experimental): Recommended servings of dairy products per day
  Interventions: Dietary Supplement: Dairy Products
- Low dairy diet (Experimental): One or fewer dairy servings per day
  Interventions: Dietary Supplement: Dairy Servings

INTERVENTIONS:
Dietary Supplement: Dairy Products — See the effect dairy product has on fat oxidation in overweight individuals expending the same amount of energy
  Other Names: Recommended dairy servings per day
  Arms: Recommended dairy diet
Dietary Supplement: Dairy Servings — Continue baseline consumption of one or fewer servings of dairy per day
  Other Names: One or fewer servings of dairy per day
  Arms: Low dairy diet

SUMMARY:
The investigators propose a randomized trial comparing higher levels of dairy intake compared to lower levels of dairy intake. Participants will be 20 boys and girls, age 10-13, overweight (>85%) who are currently consuming 1 or fewer servings of dairy per day. Each participant will be randomized to either higher or lower levels of dairy intake. A baseline calorimeter stay will determine 24-hour energy needs. Participants will then receive the diet they have been randomized to receive for 6 days and will then have a second calorimeter stay. During this 2nd stay, each participant will continue to receive the diet they were randomized to receive and will achieve a 300 kcal energy deficit through physical activity. The investigators hypothesize that children who receive a 300 kcal energy deficit from the energy expenditure of exercise and receive 3 to 4 servings of dairy products will show greater increases in fat oxidation compared to children who receive a 300 kcal energy expenditure of exercise and receive 1 or fewer servings of dairy products.

DETAILED DESCRIPTION:
The study objective was to conduct a randomized clinical trial comparing enhanced levels of dairy consumption to lower levels of dairy consumption during an energy deficit resulting from 300 kcal of exercise. Participants were 24 sedentary and overweight boys, 13-15 years of age and girls, 12 to 14 years of age, and consuming 1 or fewer servings of dairy and less than 600 mg calcium per day at baseline. Participants were randomly assigned to either higher or lower dairy for 6 days and then crossed over to the opposite treatment subsequent to 2 weeks of wash out. The investigators provided all meals and snacks for the participants during the higher and lower dairy conditions. During the wash out period, participants were instructed to consume their normal diet as assessed at baseline which consisted of 1 or fewer servings of dairy and less than 600 mg calcium. Participants stayed in the calorimeter at baseline, day 7, and day 28 (end of study), after crossover. The calorimeter measured substrate oxidation under the condition of a 300 kcal energy deficit due to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Must be overweight
* and 10-13 years old
* currently consuming 1 or fewer servings of dairy
* less than 600 mg calcium per day

Exclusion Criteria:

* not meeting the above criteria
* must be present for duration of the study

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
24hr fat oxidation | 24 hrs
  Fat oxidation over a 24 hr period will be measured using whole room indirect calorimetry.

SECONDARY OUTCOMES:
24hr energy expenditure | baseline, 7 days after each diet
  Energy Expenditure over a 24 hr period will be measured using whole room indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Donnelly, EdD, Principal Investigator — Univesity of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States